CLINICAL TRIAL: NCT05013008
Title: A Non-blinded Retrospective Biomarker add-on Study to FIGARO-DKD for Bioprofiling the Pharmacodynamic Response to Finerenone in FIGARO-DKD Subjects
Brief Title: An add-on Study to the FIGARO-DKD Study Called FIGARO-BM to Learn About the Link Between Biomarkers (Substances in the Blood Used as Indicators of Biological Processes, Disease Processes or Responses to Medication) and Finerenone in FIGARO-DKD Participants
Acronym: FIGARO-BM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21952; 2021-003053-37 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-08-19 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Experimental): Participants received finerenone 10 mg or 20 mg once daily in addition to standard of care therapy in previous interventional Phase 3 trial FIGARO-DKD. No new intervention was administered in this biomarker study.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)
- Placebo (Placebo Comparator): Participants received matching placebo once daily in addition to standard of care therapy in previous interventional Phase 3 trial FIGARO-DKD. No new intervention was administered in this biomarker study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Oral tablet; starting at 10 mg or 20 mg; once daily; received in previous interventional Phase 3 trial FIGARO-DKD; no new intervention was administered in this biomarker study.
  Arms: Finerenone
Drug: Placebo — Oral tablet; starting at 10 mg or 20 mg; once daily; received in previous interventional Phase 3 trial FIGARO-DKD; no new intervention was administered in this biomarker study.
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD), a long-term, progressive decrease in the kidneys' ability to work properly. When CKD happens in people with type 2 diabetes mellitus, a condition characterized by high blood sugar levels, CKD is also referred to as diabetic kidney disease (DKD).

FIGARO-BM is an add-on study in which blood draws that were collected in the FIGARO-DKD study are further analyzed. No additional blood draws (also referred to as biological samples) or data will be obtained from the participants, nor will any additional or new study intervention be introduced. No visit or patient contact other than for obtaining the agreement by the patients (also called informed consent) will be required.

Inflammation and scarring are both seen as responsible for worsening of chronic kidney disease. There is much information from animal studies that the study treatment finerenone (BAY94-8862) works against inflammation and against scarring (also called fibrosis) in organs such as the kidney.

In this exploratory study researchers want to learn more about the study treatment finerenone (BAY94-8862). To find this out, this study will examine substances called biomarkers in blood draws from participants in the FIGARO-DKD study. Biomarkers are used as indicators of biological processes, disease processes or responses to medication. The biomarkers that will be examined stand for inflammation, organ scarring (also called fibrosis), blood vessel function and congestion.

The main question of this study is whether there are differences between these biomarkers in the group of participants who received finerenone and the group of participants who received a placebo in the FIGARO-DKD study. A placebo looks like a treatment but does not have any medicine in it. To answer this question, the researchers will compare the levels of these biomarkers between the two groups at different time points after starting the study treatment. Blood samples for this study will be obtained from FIGARO-DKD study sites with a high number of participants who had been treated with finerenone or placebo for at least 24 months. This information will be combined with other information from biomarker examinations already available in the FIGARO-DKD study.

ELIGIBILITY:
Inclusion Criteria:

* This study will only include participants who were enrolled in the FIGARO-DKD study (NCT02545049) and had received up to 20 mg finerenone or placebo for ≥24 months.
* For each participant, pharmacokinetic (PK) plasma samples from Visit 3 and at least 2 other Visits (Visit 5, Visit 8, Visit 11) must be available on storage from the main study FIGARO-DKD.

Exclusion Criteria:

* Participants which did not show overall compliance of 80 to 120% with study intervention in FIGARO-DKD.
* Participants which were not part of the full analysis set (FAS) of FIGARO-DKD.
* Participants with known fatal outcome.
* Participants with baseline estimated glomerular filtration rate (eGFR) ≤25 mL/min/1.73m^2.
* Participants with low baseline risk (normal albuminuria and eGFR≥60 mL/min/1.73m^2).
* Sponsor request (after discussion with the investigator), for reasons such as a significant protocol deviation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (115):
- United States (13):
  - Valley Clinical Trials, Inc. - Northridge, Northridge, California
  - Saviers Medical Group, Port Hueneme, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Florida Kidney Physicians - Fort Lauderdale, Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Randolph Medical Associates, Asheboro, North Carolina
  - Clinical Advancement Center, PLLC, San Antonio, Texas
- Australia (2):
  - Illawarra Diabetes Service, Wollongong, New South Wales
  - Melbourne Renal Research Group, Reservoir, Victoria
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Klinik Landstraße - Krankenhaus Rudolfstiftung, Vienna
  - Zentrum f. klinische Studien Dr. Hanusch GmbH, Vienna
- Belgium (2):
  - UZ Gent, Ghent
  - AZ Delta, Roeselaere
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment St. Ivan Rilski - Gorna Oryahovitsa | Nephrology Department, Gorna Oryahovitsa
  - DCC 2 - Plovdiv EOOD, Plovdiv
  - MHAT Sveti Pantaleymon - Yambol, Yambol
- Canada (4):
  - Fraser Clinical Trials, Inc., New Westminster, British Columbia
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Manna Research (Mirabel), Mirabel, Quebec
  - Clinique des Maladies Lipidques de Quebec, Québec
- Nefrologicka ambulance, Prague, Czechia
- Denmark (9):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Sydvestjysk Sygehus Esbjerg, Endocrinology dept., Esbjerg
  - Capital Region | Gentofte Hospital - Cardiology Research, Hellerup
  - Herlev Hospital - Endocrinology dept., Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Holbæk Sygehus, Holbæk
  - Holstebro Hospital, Endocrinology dept., Holstebro
  - Bispebjerg Hospital, København NV
  - Viborg Sygehus, Viborg
- Finland (3):
  - Terveystalo Oulu, Oulu
  - Lääkärikeskus Minerva, Rauma
  - Turun yliopistollinen keskussairaala, Turku
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital Hong Kong, Shatin
  - Tung Wah Hospital, Sheung Wan
- Israel (7):
  - Barzilai Medical Center | Nephrology & Hypertension Dept., Ashkelon
  - Edith Wolfson Medical Center, Holon
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Nazareth Trust Hospital EMMS, Nazareth
  - Clalit Health Services, Midgal Hamea, Tel Aviv
  - DMC - Diabetes Medical Center, Tel Aviv
- Italy (4):
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - Istituto Ricerche Farmacologiche Mario Negri IRCCS, Bergamo, Lombardy
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Santi Paolo e Carlo, Milan, Lombardy
- Japan (22):
  - Kohnodai Hospital, NC for Global Health and Medicine, Ichikawa, Chiba
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Shirakawa Kosei General Hospital, Shirakawa, Fukushima
  - Higashihiroshima Medical Center, Higashihiroshima, Hiroshima
  - Jiyugaoka YAMADA Clinic, Obihiro, Hokkaido
  - Nakakinen Clinic, Naka, Ibaraki
  - Noritake Clinic, Ushiku, Ibaraki
  - Komatsu Municipal Hospital, Komatsu, Ishikawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - Sugiura Clinic, Kawaguchi, Saitama
  - Association of healthcare corporation, Oyama East Clinic, Oyama, Tochigi
  - Fukuoka University Hospital, Fukuoka
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Kyosokai AMC NISHI-UMEDA Clinic, Osaka
  - Kitano Hospital, Osaka
- Albert Schweitzer Ziekenhuis, locatie Zwijndrecht, Zwijndrecht, Netherlands
- Centro Clinico Academico - Braga, Braga, Portugal
- Russia (14):
  - First City Clinical Hospital n.a. E.E. Volosevich, Arkhangelsk
  - Izhevsk City Clinical Hospital #9, Izhevsk
  - Sci-Res. Institute of Complex Cardiovascular Disorders, Kemerovo
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Center of cardiology and neurology, Kirov
  - Regional Clinical Hospital #1 n.a. prof. S.V. Ochapovsky, Krasnodar
  - Moscow State University n.a. M.V. Lomonosov, Moscow
  - Moscow State Univ. of Med. & Stomatology n.a. A.I. Evdokimov, Moscow
  - PHI "Central Clinical Hospital "RZD-Medicine", Moscow
  - City Clinical Hospital #13 Nizhny Novgorod, Nizhny Novgorod
  - Saratov City Clinical Hospital #9, Saratov
  - Voronezh Regional Clinical Consultancy-Diagnostic Center, Voronezh
  - City Outpatient Clinic #4, Voronezh
  - Clinical Hospital for Emergency Care n.a. N.V.Solovyov, Yaroslavl
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- South Korea (7):
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gang''weondo
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Gerencia de Gestion Integrada A Coruna | Department of Endocrinology and Nutrition, A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Lugar Da Pega, A Coruña
  - Hospital SAS de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital del Mar | Nephrology Department, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (3):
  - PTC-Primary care Trial Center, Gothenburg
  - Avdelningen för kliniska prövningar AKP, Örebro
  - ClinSmart, Uppsala
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Far Eastern Memorial Hospital | Nephrology Department, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21952
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 21 countries/regions between 18 August 2021 (first subject first visit) and 31 December 2021 (last subject last visit).
Pre-assignment Details: Overall, 952 participants from previous FIGARO-DKD study (NCT02545049) were screened for this FIGAGRO-BM study. Of the 952 screened (i.e. signed informed consent available either for this FIGARO-BM study or for the protocol addendum for FIGARO-DKD), 1 participant was a screening failure and 30 participants missed treatment and/or biomarker data at Visit 3 or 11 in FIGARO-DKD. The remaining 921 participants were included in the modified biomarker full analysis set of FIGAGRO-BM study.
Period: Overall Study
Arm/Group | Finerenone | Placebo
Started | 483 | 468
mBFAS (Modified biomarker full analysis set (mBFAS)) | 478 | 443
Completed | 478 | 443
Not Completed | 5 | 25
Not completed — Exclusion from mBFAS | 5 | 25

BASELINE CHARACTERISTICS:
Population: Modified biomarker full analysis set (mBFAS): All participants with valid informed consent for this biomarker study, which met the following criteria: a. Study enrollment criteria as defined in the study protocol. b. Analyzed biomarker samples at Visit 3 (4 months) and Visit 11 (36 months); Biomarker samples that were shipped at ambient temperatures were not analyzed. c. On Treatment at Visit 3 and Visit 11.
Groups:
- Total: Total of all reporting groups
Arm/Group | Finerenone | Placebo | Total
Number analyzed (Participants) | 478 | 443 | 921
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.55 (9.50) | 64.15 (9.65) | 63.84 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 112 | 232
  Male | 358 | 331 | 689
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 173 | 151 | 324
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 7 | 15
  White | 293 | 283 | 576
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 2
Plasma biomarker levels after 4 months of treatment [Geometric Mean (Standard Deviation); unit: Linear NPX (2^NPX)] — The normalized protein expression (NPX) of biomarker levels were analyzed for the set of 27 pre-defined plasma biomarkers. NPX is a unit on log2-scale that is logarithmically related to protein concentration. Linear NPX (2^NPX) was calculated for descriptive analyses of the biomarker levels at each visit. Visit 3 (4 months of treatment) data were considered as baseline for the biomarker measurements as no pre-dose samples were available from FIGARO-DKD. Population: Participants in mBFAS with available data for each biomarker measurement
  Linear NPX (2^NPX)
    Matrilysin (P09237): number analyzed (Participants) | 427 | 403 | 830
    Matrilysin (P09237) | 19.618 (1.148) | 18.956 (1.203) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    von Willebrand factor (P04275): number analyzed (Participants) | 472 | 434 | 906
    von Willebrand factor (P04275) | 3.200 (1.793) | 2.338 (1.629) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    CCN family member 4 (O95388): number analyzed (Participants) | 470 | 436 | 906
    CCN family member 4 (O95388) | 1.600 (1.337) | 1.578 (1.374) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Transforming growth factor beta-1 proprotein (P01137): number analyzed (Participants) | 471 | 436 | 907
    Transforming growth factor beta-1 proprotein (P01137) | 1.480 (1.327) | 1.425 (1.349) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Transforming growth factor beta receptor type 3 (Q03167): number analyzed (Participants) | 472 | 434 | 906
    Transforming growth factor beta receptor type 3 (Q03167) | 1.583 (1.631) | 1.776 (1.624) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Interleukin-15 receptor subunit alpha (Q13261): number analyzed (Participants) | 435 | 408 | 843
    Interleukin-15 receptor subunit alpha (Q13261) | 1.678 (1.432) | 1.614 (1.450) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Metalloproteinase inhibitor 1 (P01033): number analyzed (Participants) | 432 | 408 | 840
    Metalloproteinase inhibitor 1 (P01033) | 1.818 (1.450) | 1.824 (1.349) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Pappalysin-1 (Q13219): number analyzed (Participants) | 435 | 408 | 843
    Pappalysin-1 (Q13219) | 0.171 (3.066) | 0.164 (2.762) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Proto-oncogene tyrosine-protein kinase Src (P12931): number analyzed (Participants) | 471 | 438 | 909
    Proto-oncogene tyrosine-protein kinase Src (P12931) | 1.770 (2.614) | 1.535 (2.229) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Protein AMBP (P02760): number analyzed (Participants) | 470 | 436 | 906
    Protein AMBP (P02760) | 1.595 (1.226) | 1.611 (1.225) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Uromodulin (P07911): number analyzed (Participants) | 443 | 405 | 848
    Uromodulin (P07911) | 0.582 (1.752) | 0.699 (1.531) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Aminopeptidase N (P15144): number analyzed (Participants) | 461 | 433 | 894
    Aminopeptidase N (P15144) | 1.224 (1.273) | 1.248 (1.300) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Tumor necrosis factor receptor superfamily member 1A (P19438): number analyzed (Participants) | 476 | 441 | 917
    Tumor necrosis factor receptor superfamily member 1A (P19438) | 2.105 (1.606) | 2.107 (1.575) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Plasminogen activator inhibitor 1 (P05121): number analyzed (Participants) | 472 | 434 | 906
    Plasminogen activator inhibitor 1 (P05121) | 1.349 (2.148) | 1.261 (1.868) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    CCN family member 2 (P29279): number analyzed (Participants) | 473 | 439 | 912
    CCN family member 2 (P29279) | 1.245 (1.585) | 1.258 (1.360) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Urokinase plasminogen activator surface receptor (Q03405): number analyzed (Participants) | 473 | 439 | 912
    Urokinase plasminogen activator surface receptor (Q03405) | 1.744 (1.699) | 1.725 (1.398) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    C-C motif chemokine 14 (Q16627): number analyzed (Participants) | 472 | 441 | 913
    C-C motif chemokine 14 (Q16627) | 3.013 (1.667) | 3.056 (1.426) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    C-C motif chemokine 16 (O15467): number analyzed (Participants) | 472 | 434 | 906
    C-C motif chemokine 16 (O15467) | 1.625 (1.776) | 1.633 (1.637) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Collagen alpha-1(I) chain (P02452): number analyzed (Participants) | 472 | 434 | 906
    Collagen alpha-1(I) chain (P02452) | 0.646 (1.675) | 0.693 (1.497) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Decorin (P07585): number analyzed (Participants) | 427 | 403 | 830
    Decorin (P07585) | 1.523 (1.233) | 1.526 (1.233) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    C-C motif chemokine 2 (P13500): number analyzed (Participants) | 444 | 407 | 851
    C-C motif chemokine 2 (P13500) | 3.065 (1.285) | 3.209 (1.367) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Matrix metalloproteinase-9 (P14780): number analyzed (Participants) | 476 | 441 | 917
    Matrix metalloproteinase-9 (P14780) | 1.329 (2.202) | 1.176 (1.985) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    E-selectin (P16581): number analyzed (Participants) | 472 | 434 | 906
    E-selectin (P16581) | 1.235 (1.828) | 1.200 (1.577) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Thrombospondin-2 (P35442): number analyzed (Participants) | 476 | 441 | 917
    Thrombospondin-2 (P35442) | 1.421 (1.655) | 1.452 (1.649) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Retinoic acid receptor responder protein 2 (Q99969): number analyzed (Participants) | 472 | 441 | 913
    Retinoic acid receptor responder protein 2 (Q99969) | 2.201 (1.580) | 2.252 (1.418) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    C-X-C motif chemokine 16 (Q9H2A7): number analyzed (Participants) | 472 | 434 | 906
    C-X-C motif chemokine 16 (Q9H2A7) | 1.341 (1.586) | 1.353 (1.338) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.
    Dickkopf-related protein 3 (Q9UBP4): number analyzed (Participants) | 472 | 434 | 906
    Dickkopf-related protein 3 (Q9UBP4) | 1.827 (1.541) | 1.925 (1.460) | NA (NA) — Biomarker data at Visit 3 were considered as baseline as pre-dose samples were not available. The study objective was to analyze the change in biomarker levels after 36 months (Visit 11) vs. 4 months (Visit 3) of treatment of participants in each arm. The analysis focused on the change over time per biomarker and per treatment and a display of total was not considered appropriate for the absolute biomarker levels, as an effect of the treatment within the first 4 month cannot fully be excluded.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Plasma Biomarker Levels After 36 Months of Treatment Versus 4 Months of Treatment in a Set of 27 Pre-defined Biomarkers
Description: The normalized protein expression (NPX) of biomarker levels were analyzed for the set of 27 pre-defined plasma biomarkers. NPX is a unit on log2-scale that is logarithmically related to protein concentration. Linear NPX (2^NPX) was calcuated for descriptive analyses of the biomarker levels at each visit. Ratios of Visit 11 (36 months of treatment) to Visit 3 (4 months of treatment) were calculated to show the change in the plasma biomarker levels. Visit 3 (4 months of treatment) data were considered as baseline for the biomarker measurements as no pre-dose samples were available from FIGARO-DKD. Note, NPX units (Olink concentration units) are always relative units and can only be interpreted in the context of an individual study, i.e. to compare two conditions or timepoints ("change in NPX"). Equal nominal concentration values (same NPX units) for two different biomarkers measured by Olink Explore does not mean that both markers have the same absolute concentration.
Time Frame: At 4 months (Visit 3) of treatment and 36 months (Visit 11) of treatment
Population: Participants in mBFAS with available data for each biomarker measurement
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 478 | 443
Ratio
  Matrilysin (P09237): number analyzed (Participants) | 387 | 386
  Matrilysin (P09237) | 1.014 (1.125) | 1.062 (1.201)
  von Willebrand factor (P04275): number analyzed (Participants) | 466 | 429
  von Willebrand factor (P04275) | 0.979 (1.773) | 1.131 (1.765)
  CCN family member 4 (O95388): number analyzed (Participants) | 461 | 433
  CCN family member 4 (O95388) | 1.109 (1.266) | 1.164 (1.329)
  Transforming growth factor beta-1 proprotein (P01137): number analyzed (Participants) | 463 | 433
  Transforming growth factor beta-1 proprotein (P01137) | 1.122 (1.312) | 1.184 (1.369)
  Transforming growth factor beta receptor type 3 (Q03167): number analyzed (Participants) | 466 | 429
  Transforming growth factor beta receptor type 3 (Q03167) | 1.133 (1.687) | 1.224 (1.649)
  Interleukin-15 receptor subunit alpha (Q13261): number analyzed (Participants) | 410 | 382
  Interleukin-15 receptor subunit alpha (Q13261) | 1.121 (1.402) | 1.179 (1.442)
  Metalloproteinase inhibitor 1 (P01033): number analyzed (Participants) | 425 | 402
  Metalloproteinase inhibitor 1 (P01033) | 1.056 (1.456) | 1.105 (1.381)
  Pappalysin-1 (Q13219): number analyzed (Participants) | 410 | 382
  Pappalysin-1 (Q13219) | 1.088 (3.371) | 1.273 (3.034)
  Proto-oncogene tyrosine-protein kinase Src (P12931): number analyzed (Participants) | 466 | 434
  Proto-oncogene tyrosine-protein kinase Src (P12931) | 0.926 (2.902) | 1.000 (2.492)
  Protein AMBP (P02760): number analyzed (Participants) | 461 | 433
  Protein AMBP (P02760) | 1.034 (1.168) | 1.045 (1.166)
  Uromodulin (P07911): number analyzed (Participants) | 437 | 400
  Uromodulin (P07911) | 0.980 (1.513) | 0.956 (1.388)
  Aminopeptidase N (P15144): number analyzed (Participants) | 453 | 427
  Aminopeptidase N (P15144) | 1.005 (1.263) | 1.020 (1.316)
  Tumor necrosis factor receptor superfamily member 1A (P19438): number analyzed (Participants) | 470 | 436
  Tumor necrosis factor receptor superfamily member 1A (P19438) | 1.151 (1.506) | 1.184 (1.516)
  Plasminogen activator inhibitor 1 (P05121): number analyzed (Participants) | 466 | 429
  Plasminogen activator inhibitor 1 (P05121) | 0.945 (2.089) | 0.972 (1.909)
  CCN family member 2 (P29279): number analyzed (Participants) | 470 | 433
  CCN family member 2 (P29279) | 1.083 (1.548) | 1.103 (1.395)
  Urokinase plasminogen activator surface receptor (Q03405): number analyzed (Participants) | 470 | 433
  Urokinase plasminogen activator surface receptor (Q03405) | 1.109 (1.661) | 1.127 (1.379)
  C-C motif chemokine 14 (Q16627): number analyzed (Participants) | 464 | 435
  C-C motif chemokine 14 (Q16627) | 1.072 (1.617) | 1.092 (1.401)
  C-C motif chemokine 16 (O15467): number analyzed (Participants) | 466 | 429
  C-C motif chemokine 16 (O15467) | 1.044 (1.607) | 1.055 (1.416)
  Collagen alpha-1(I) chain (P02452): number analyzed (Participants) | 466 | 429
  Collagen alpha-1(I) chain (P02452) | 1.101 (1.680) | 1.112 (1.534)
  Decorin (P07585): number analyzed (Participants) | 387 | 386
  Decorin (P07585) | 1.086 (1.202) | 1.088 (1.250)
  C-C motif chemokine 2 (P13500): number analyzed (Participants) | 426 | 386
  C-C motif chemokine 2 (P13500) | 1.001 (1.329) | 1.003 (1.409)
  Matrix metalloproteinase-9 (P14780): number analyzed (Participants) | 470 | 436
  Matrix metalloproteinase-9 (P14780) | 1.074 (2.303) | 1.080 (2.108)
  E-selectin (P16581): number analyzed (Participants) | 466 | 429
  E-selectin (P16581) | 1.009 (1.681) | 1.010 (1.432)
  Thrombospondin-2 (P35442): number analyzed (Participants) | 470 | 436
  Thrombospondin-2 (P35442) | 1.054 (1.533) | 1.056 (1.533)
  Retinoic acid receptor responder protein 2 (Q99969): number analyzed (Participants) | 464 | 435
  Retinoic acid receptor responder protein 2 (Q99969) | 1.035 (1.569) | 1.022 (1.517)
  C-X-C motif chemokine 16 (Q9H2A7): number analyzed (Participants) | 466 | 429
  C-X-C motif chemokine 16 (Q9H2A7) | 1.058 (1.562) | 1.063 (1.330)
  Dickkopf-related protein 3 (Q9UBP4): number analyzed (Participants) | 466 | 429
  Dickkopf-related protein 3 (Q9UBP4) | 1.050 (1.452) | 1.055 (1.427)
Statistical Analysis 1: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Matrilysin (P09237) was analyzed; Test type: Other — The hypotheses 'H0i: βi=0' (i=1,…,27) were tested at a two-sided significance level of 5%, where βi was the estimator for the difference in log-transformed ratios of biomarker levels of Visit 11 to Visit 3 between finerenone and placebo group for the i-th of the 27 pre-specified biomarkers; p = 0.001, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 2: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of von Willebrand factor (P04275) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 3: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of CCN family member 4 (O95388) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.044, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 4: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of TGF beta-1 proprotein (P01137) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.044, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 5: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of TGF beta receptor type 3 (Q03167) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.127, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 6: Comparison: Finerenone vs Placebo; The NPX differences (corresponding to log-transformed ratio to baseline) of IL-15 receptor subunit alpha (Q13261) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.210, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 7: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Metalloproteinase inhibitor 1 (P01033) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.215, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 8: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Pappalysin-1 (Q13219) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.215, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 9: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Proto-oncogene c-Src (P12931) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.745, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 10: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Protein AMBP (P02760) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.762, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 11: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Uromodulin (P07911) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.762, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 12: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Aminopeptidase N (P15144) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.762, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 13: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of TNFRSF1A (P19438) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.762, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 14: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Plasminogen activator inhibitor 1 (P05121) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.917, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 15: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of CCN family member 2 (P29279) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.917, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 16: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of uPAR (Q03405) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.917, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 17: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of C-C motif chemokine 14 (Q16627) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.917, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 18: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of C-C motif chemokine 16 (O15467) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 19: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Collagen alpha-1(I) chain (P02452) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 20: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Decorin (P07585) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 21: Comparison: Finerenone vs Placebo; The NPX differences (corresponding to log-transformed ratio to baseline) of C-C motif chemokine 2 (P13500) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 22: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Matrix metalloproteinase-9 (P14780) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 23: Comparison: Finerenone vs Placebo; The NPX differences (corresponding to log-transformed ratio to baseline) of E-selectin (P16581) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 24: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Thrombospondin-2 (P35442) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 25: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of RARRES2 (Q99969) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 26: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of C-X-C motif chemokine 16 (Q9H2A7) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value
Statistical Analysis 27: Comparison: Finerenone vs Placebo; The NPX difference (corresponding to log-transformed ratio to baseline) of Dickkopf-related protein 3 (Q9UBP4) was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.979, t-test, 2 sided — Benjamini-Hochberg adjusted P-value was calculated using the log2-scaled NPX value

ADVERSE EVENTS:
Description: This study was a retrospective, add-on biomarker study to the multi-center, interventional Phase 3 study FIGARO-DKD (NCT02545049). There was no study-specific safety assessments in this study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed therefore total number of participants at risk is "0" . Safety of the subjects was monitored within the FIGARO-DKD study.
Arm/Group | Finerenone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was a retrospective, add-on study to the multi-center, interventional Phase 3 study FIGARO-DKD (NCT02545049). Blood plasma samples that were originally collected for PK analysis during the conduct of FIGARO-DKD study. Visit 3 (4 months of treatment) data were considered as baseline for the biomarker measurements as no pre-dose samples were available from FIGARO-DKD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT05013008/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT05013008/SAP_001.pdf